CLINICAL TRIAL: NCT01014065
Title: A Prospective Study of Acute Cardiovascular Effects of First-line Sunitinib in Metastatic Renal Cell Carcinoma Patients
Brief Title: A Prospective Study of Acute Cardiovascular Effects of First-line Sunitinib in Metastatic Renal Cell Carcinoma Patients (SUnitinib Prospective CardiovasculaR Effect)
Acronym: SUPER
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 00028 / 24942
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Renal Cell Carcinoma; Cardiotoxicity; Heart Failure; Hypertension
Keywords: sunitinib; cardiac MRI; maximal exercise testing; biomarkers; pharmacokinetics
MeSH Terms: conditions — Carcinoma, Renal Cell; Cardiotoxicity; Heart Failure; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine banked
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with renal cell carcinoma scheduled to receive sunitinib

SUMMARY:
While sunitinib can be very helpful to treat kidney cancer, these medications can also cause side effects, including heart damage. Studies performed in the past did not look at heart function in detail, so the investigators do not know what happens to the heart when people start sunitinib treatment. The aim of the study is to prospectively study acute effects of sunitinib on heart function, overall fitness and blood markers of heart disease.

DETAILED DESCRIPTION:
Participants will undergo cardiac MRI, maximal exercise testing(VO2 peak), blood and urine samples before and after 2 treatments of sunitinib. An extra blood sample will be collected the 2nd week of the first treatment to check blood levels of sunitinib. We will also examine routine CT scans to study body composition.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of metastatic renal cell carcinoma
* Eligible to receive first-line sunitinib
* Willingness to attend Cross Cancer Institute and University of Alberta for study-related assessments
* Karnofsky Performance Status (KPS)82 ≥ 70
* Age ≥ 18 years of age
* Adequate creatinine clearance to receive gadolinium
* All patients with bone metastases are eligible; those with lesions identified at weight-bearing bones will undergo plain films to evaluate fracture risk prior to CPET;
* Fluent in English language
* No contraindication to MRI or other concern eg., metallic implants, claustrophobia

Exclusion Criteria:

* Prior systemic therapy for mRCC
* Documented history of major cardiac event in last year i.e. MI, unstable angina, CABG, symptomatic CHF, CVA or TIA, or pulmonary embolism
* Pregnancy
* Other severe condition or abnormality that, in the judgement of the investigator or treating oncologist, would make participation in this study inappropriate
* Unstable brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal cell carcinoma scheduled to receive sunitinub.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haykowsky, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada